CLINICAL TRIAL: NCT05185947
Title: Phase II Study of Intravenous and Intraperitoneal Paclitaxel and Oral Nilotinib for Peritoneal Carcinomatosis From Colorectal, Appendiceal, Small Bowel, Gastric, Cholangiocarcinoma, Breast, Ovarian, or Other Gynecologic Primary Cancer
Brief Title: Study of Intravenous and Intraperitoneal Paclitaxel and Oral Nilotinib for Peritoneal Carcinomatosis From Colorectal, Appendiceal, Small Bowel, Gastric, Cholangiocarcinoma, Breast, Ovarian, or Other Gynecologic Primary Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000237; 000237-C
Record Dates: First submitted 2022-01-08; First posted 2022-01-11 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03-05

CONDITIONS: Gynecologic Cancer; Gynecologic Neoplasms; Peritoneal Carcinomatosis; Peritoneal Neoplasms; Ovarian Cancer; Ovarian Neoplasms; Colorectal Cancer; Colorectal Neoplasms; Appendiceal Cancer; Appendiceal Neoplasms
Keywords: Taxol; Tasigna; Peritoneal Carcinomatosis Index (PCI); cytoreductive surgery (CRS); Unresectable; SMART System; necrosis; Ki-67; Peritoneal Metastasis; Progression Free Survival
MeSH Terms: conditions — Genital Neoplasms, Female; Peritoneal Neoplasms; Ovarian Neoplasms; Colorectal Neoplasms; Appendiceal Neoplasms; Necrosis | interventions — Paclitaxel; nilotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/ IP Catheter Placement and Bidirectional Chemotherapy (Experimental): IP and IV paclitaxel administration with oral nilotinib
  Interventions: Drug: Paclitaxel; Drug: Nilotinib

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel: Intraperitoneal (IP) paclitaxel will be dosed at 60 mg/m2 to be infused over 1 hour on Day 1 of each 3-week cycle; participants with unresectable, but stable or responding disease after C1 through C3 will dose increase IP paclitaxel to 80 mg/m2 for Cycles 4-6. Intravenous (IV) paclitaxel will be infused over 1 hour on Day 2 of the first week of Cycle 1, followed by Day 1 of the subsequent treatment weeks; IV paclitaxel will be dosed at 60 mg/m2 for Week 1 of Cycle 1 and, if tolerated, at 80 mg/m2 for subsequent treatments.
Drug: Nilotinib — Oral nilotinib will be dosed at 300 mg twice daily. Nilotinib will be administered continually from the loading dose (Day -4) leading up to laparoscopy #2 onward.

SUMMARY:
Background:

Tumors that have spread to the lining of the abdomen from other cancers, such as cancer of the appendix, colon, or ovary, are called peritoneal carcinomatosis. In most cases, outcomes are poor. Researchers want to test a new treatment.

Objective:

To learn if the combination of oral nilotinib plus paclitaxel given by IV and directly into the abdomen can reduce tumors enough for people to have surgery.

Eligibility:

Adults aged 18 and older with peritoneal carcinomatosis that is too widespread for surgery.

Design:

Participants will be screened with:

Physical exam

Medical history

Blood and urine tests

Electrocardiogram

Laparoscopy. They will get general anesthesia. Small cuts will be made in their abdomen. Tissue and fluid samples will be taken.

Surveys about their health

CT scans of their torso

Participants will have up to 4 more laparoscopies. During the first procedure, a port will be placed under the skin of their abdomen (an IP port). It will be attached to a catheter that is placed in their abdomen.

Participants will get treatment in 3-week cycles, for 3 or 6 cycles. They will take nilotinib by mouth twice daily. They will get paclitaxel by IP port (once per cycle) and by IV (twice per cycle). After cycles 3 and 6, they will have a laparoscopy and CT scans. Then they may take nilotinib and get IV paclitaxel for up to 1 year.

At study visits, participants will repeat some screening tests.

About 6 weeks after treatment ends and then every 3 months for 3 years, participants will have follow-up visits at NIH or with their local doctor.

DETAILED DESCRIPTION:
Background:

* Peritoneal carcinomatosis is uniformly fatal if untreated; despite advances in systemic chemotherapy, cytoreductive surgery, and intraperitoneal chemotherapy, survival remains poor for the majority of patients
* The combination of oral nilotinib and intravenous paclitaxel has demonstrated pre-clinical and clinical synergism in the treatment of solid tumors, with an ongoing Phase I trial at the NIH
* The synergy of oral nilotinib with intraperitoneal paclitaxel remains to be characterized
* This study involves the combination of intravenous and intraperitoneal paclitaxel and oral nilotinib for unresectable peritoneal carcinomatosis from colorectal, appendiceal, small bowel, gastric, cholangiocarcinoma, breast, ovarian, or other gynecologic primary histologies

Objective:

-To evaluate efficacy of bidirectional chemotherapy using intraperitoneal and intravenous paclitaxel and oral nilotinib by calculating the rate of downstaging of peritoneal disease burden to become resectable, based on Peritoneal Carcinomatosis Index (PCI)

Eligibility:

* Participants >= 18 years of age with histologically confirmed peritoneal carcinomatosis of colorectal, appendiceal, small bowel, gastric, cholangiocarcinoma, breast, ovarian, or other gynecologic primary histology
* Demonstrated resistance or lack of response to at least one line of already approved and available systemic chemotherapy
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to study drugs
* No intraperitoneal chemotherapy within the last six months
* Deemed unable to undergo complete cytoreduction

Design:

* Phase II open-label, non-randomized study
* After confirmation of eligibility, at the time of diagnostic laparoscopy, biopsies will be taken, and an intraperitoneal catheter will be placed for subsequent chemotherapy administration
* Up to 6 cycles will be planned, with restaging laparoscopy and biopsies after Cycles 3 and 6

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria.

* Histological confirmation of peritoneal carcinomatosis from colorectal, appendiceal, small bowel, gastric, cholangiocarcinoma, breast, ovarian, or other gynecologic (i.e., endometrial, fallopian tube, primary peritoneal, cervical) primary by the Laboratory of Pathology, NCI.
* Participants must have been treated with at least one line of approved systemic chemotherapy, with demonstrated resistance or lack of response
* Measurable or evaluable disease as defined by RECIST v1.1. criteria and/or by Peritoneal Carcinomatosis Index (PCI)
* Participants must be assessed to not be candidates for cytoreductive surgery, with laparoscopically assessed PCI score thresholds as indicated below:

  --Primary Histology PCI Cutoff for Eligibility
  * Gastric Total Score >= 10 (out of 39 possible points)
  * Others Total Score >= 20 (out of 39 possible points)
  * Any Jejunoileal Score >= 4 (out of 12 possible points)
* Age >= 18 years
* ECOG performance status <= 2 (Karnofsky >= 60%).
* Participants must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count >= 1,000/mcL
  * Platelets >= 100,000/mcL
  * Total bilirubin within <= 1.5x institutional upper limit of normal (ULN)
  * AST (SGOT)/ ALT (SGPT) <= 3x institutional ULN, or <= 5.0x ULN in participants with liver metastases (only)
  * Serum potassium and magnesium greater than institutional lower limit of normal
  * Creatinine <= 1.5 mg/dL or creatinine clearance >= 60 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal calculated using eGFR
* Nursing (including breastfeeding) participant must agree to discontinue nursing.
* Individuals of child-bearing potential (IOCBP) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 90 days after last study treatment. Should an individual of child-bearing potential suspect to be pregnant while participating in this study, the individual should inform the treating physician immediately.
* Ability of participant to understand and the willingness to sign a written informed consent document.
* Participants must agree to co-enrollment on the tissue collection protocol 13C0176, Tumor, Normal Tissue and Specimens from Patients Undergoing Evaluation or Surgical Resection of Solid Tumors

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study.

* Participants who are receiving any other investigational agents or who have received an investigational agent within 30 days prior to the start of study treatment.
* Participants with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to study drugs.
* Participants who have received systemic (i.e., oral or intravenous) chemotherapy or other anti-cancer therapy (i.e., immunotherapy) within either 5 half-lives or within 30 days of the last dose of individual agent(s) administered prior to the start of study treatment, whichever is shorter.
* Participants who have undergone major abdominal surgery within the last 12 weeks prior to the start of study treatment.

Note: Exclusion of participants who have undergone major abdominal surgery within the last 12 weeks prior to start of study treatment is to allow for scar tissue formation from that surgery to stabilize. Participant ECOG performance status will be checked to account for prolonged or difficult recoveries from other types of major surgery that would appropriately influence eligibility assessment.

* Participants who have received previous intraperitoneal chemotherapy within the last 6 months prior to the start of study treatment
* Participants requiring the use of drugs known to prolong the QT interval or known to strongly inhibit CYP3A4, 2C8. Participants on such agents at the time of screening are permitted on study if an alternative that does not have the same pharmacokinetic interactions can be found.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Note: No subject will be excluded based on a social situation prior to consultation with the Department of Social Work.
* Pregnant individuals are excluded from this study.
* Participants with HIV who have detectable viral load, or whose ART contains QTc Prolonging Medications or CYP3A4 Inhibitors regardless of viral load. (NOTE: Participants with HIV who have an undetectable viral load and have been on stable doses of ART that does not prolong the QT interval or is a strong CYP3A4, 2C8 inhibitor are eligible).
* QTcF interval of >= 450 msec at study entry, or congenital long QT syndrome.
* More than 3 liters of ascites present at initial laparoscopy, or history of more than two therapeutic paracentesis procedures, each yielding at least 1.5 liters of fluid, in the 30 days prior to initial laparoscopy, or confirmation of predominantly mucinous ascites at

the time of screening laparoscopy.

* Advanced hepatic failure, as indicated by Child-Pugh Class C cirrhosis.
* Sensory/motor neuropathy >= Grade 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-04-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate efficacy of bidirectional chemotherapy using intraperitoneal and intravenous paclitaxel and oral nilotinib by calculating the rate of downstaging of peritoneal disease burden to become resectable, based on Peritoneal Carcinomatosis Inde... | baseline, every 9 weeks during treatment, and then every 3 months for 3 years
  Rate of downstaging- i.e., the fraction of participants who are successfully downstaged to resectable based on PCI and PI discretion. The fraction of participants who are successfully down-staged to resectable by use of chemotherapy will be reported along with a 95% confidence interval.

SECONDARY OUTCOMES:
Measure overall survival (OS) and overall progression-free survival (PFS) | baseline, at peritoneal disease relapse from CR or peritoneal disease progression, or death, for up to 3 years after completion of therapy
  Kaplan-Meier method will be used; a 95% confidence interval will be reported on the median overall survival (OS) and overall progression-free survival (PFS).
Evaluate the peritoneal progression-free survival (pPFS) probability and the percentage of participants who become resectable by individual histologies | baseline, at peritoneal disease relapse from CR or peritoneal disease progression, for up to 3 years after completion of therapy
  Peritoneal progression-free survival (pPFS) probability and the percentage of participants who become resectable will be evaluated by individual histologies; median peritoneal progression-free survival (pPFS) will be reported using the Kaplan-Meier method, along with a 95% confidence interval for each histology. The fraction who are able to be down-staged to resectable will be reported for each histology along with a 95% confidence interval.
Evaluate safety and tolerability of therapy | on-going throughout treatment
  Safety will be assessed by analyzing the type, grade and frequency of toxicities in addition to laboratory data and vital signs. Adverse events (AEs) will be assessed using CTCAE v.5.0
Evaluate participants quality of life (QOL) | baseline, every 9 weeks while on treatment, then every 3 months for 3 years after completion of study therapy
  Outcomes from QOL will be reported using descriptive statistics, as well as comparing the results from before to after treatment: physical and mental health-related quality of life.
Determine peritoneal progression-free survival (pPFS) | baseline, at peritoneal disease relapse from CR or peritoneal disease progression, for up to 3 years after completion of therapy
  Kaplan-Meier method will be used to evaluate peritoneal progression-free survival (pPFS); the median peritoneal progression-free survival (pPFS) will be reported along with a 95% two-sided confidence interval, to be done for all participants.
Assess clinicopathologic response to therapy | baseline, every 9 weeks during treatment, and then every 3 months for 3 years
  Response rate by RECIST 1.1 and/or by PCI: the fractions with a clinical response will be reported for all participants along with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Blakely, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000237-C.html